CLINICAL TRIAL: NCT05469841
Title: Pupillometry and Nociception Level Index (NOL-index) for the Evaluation of Pain in Intensive Care Unit. Prospective Study in Two Centers
Brief Title: Pupillometry and Nociception Level Index for the Evaluation of Pain in Intensive Care Unit.
Acronym: NOCI-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2022-04
Record Dates: First submitted 2022-06-20; First posted 2022-07-22 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Critical Illness
Keywords: pain; intensive care; sedated; ventilated; NOL ICU; pupillometry
MeSH Terms: conditions — Critical Illness; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pupillometry (Experimental): Pain will be evaluated via pupillometry with 3 successive measurements
  Interventions: Other: Systemic pain assessment

INTERVENTIONS:
Other: Systemic pain assessment — Pain will be evaluated via i) pupillometry with 3 successive measurements ii) Behaviour Pain Scale (BPS) and Critical Care Pain Observation Tool (CPOT) score evaluated by an investigator (physician) iii) evolution of physiological parameters (ie heart rate, blood pressure, respiratory rate) iv) Nociception Level Index (NOL) index.

SUMMARY:
Pain is a frequent symptom in the intensive care unit (ICU). Critical ill patients are often intubated and sedated which makes self-evaluation of pain impossible.

Pupillary dilatation is a reflex directly related to stimuli such as pain, which can be measured by quantitative pupillometry.

Several studies in ICU showed a significant relationship between pupillary diameter variation and pain.

The nociception level index (NOL-index) is a recent noninvasive and continuous monitoring of pain essentially used in operating room.

The aim of this study is to evaluate the pupillometry and NOL index in critical ill patients in sedated patients under mechanical ventilation during the mobilization plus toilet (described in literature as not painful procedure) and tracheal suctioning (described as a painful procedure)

DETAILED DESCRIPTION:
Pain will be evaluated via i) pupillometry with 3 successive measurements ii) Behaviour Pain Scale (BPS) and Critical Care Pain Observation Tool (CPOT) score evaluated by an investigator (physician) iii) evolution of physiological parameters (ie heart rate, blood pressure, respiratory rate) iv) Nociception level index (NOL-index).

The evaluation times will be 5 minutes before care procedures (mobilization plus toilet and tracheal suctioning), during the procedures (with the worst value recorded) and 5 minutes after the procedures.

The procedures are:

* A mobilization and toilet of the patient: a priori, not a very painful procedure. The pain will be evaluated every 5 minutes during the toilet.
* Tracheal suctioning: a procedure known to be painful. The painful will be evaluated just at the end of tracheal suctioning (once the tracheal suctioning catheter is removed from the endotracheal intubation).

ELIGIBILITY:
Inclusion Criteria:

* older than18 years old
* Under invasive mechanical ventilation
* Sedated with i) a Richmond Agitation Sedation Scale (RASS) : ≥ -4 and <1, ii) being unable to evaluate their pain by a visual numeric scale

Exclusion Criteria:

* Ophthalmological diseases which could modify the pupillometric parameters
* Neurological diseases (damage of nerve III, intracranial hypertension, stroke)
* Admitted in ICU after resuscitated cardiac arrest
* Drugs that inhibit the effect of the sympathetic system (clonidine, dexmedetomidine)
* Patient under Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO)
* Patient treated by a neuromuscular blockade
* A do-not resuscitate order
* Major hemodynamic instability prohibiting planned care procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
pupillary redilatation velocity after constriction light-induced | 1 hour during procedure
  Area under the ROC curve (AUC) of pupillary re-dilation velocity measured before a potentially painful procedure to predict the occurrence of a BPS score ≥ 5 during the procedure.

SECONDARY OUTCOMES:
Nociception Level index | 1 hour during procedure
  To evaluate the predictive value of the NOL-index measured before a potentially painful procedure to predict the intensity of the pain felt during the procedure.
Systolic and diastolic Blood pressure | 1 hour during procedure
  Describe the variations of vital parameters
Heart rate | 1 hour during procedure
  Describe the variations of vital parameters
Respiratory rate | 1 hour during procedure
  Describe the variations of vital parameters
Behaviour Pain Scale | 1 hour during procedure
  Compare variations of nociception parameters during mobilizations and during tracheal aspirations Behaviour Pain Scale Score from 3 (no pain) to 12 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mai Anh NAY, MD, Study Director — Regional Hospital Center of ORLEANS
Locations (2):
- France (2):
  - Regional Hospital Center, Orléans
  - Universitary Hospital Center, Tours

IPD SHARING:
Plan to Share IPD: No